CLINICAL TRIAL: NCT05684055
Title: Community-based, eHealth Supported Management of Cardiovascular Risk Factors by Lay Village Health Workers for People With Controlled and Uncontrolled Arterial Hypertension in Rural Lesotho: Joint Protocol for Two Cluster-randomized Trials Within the ComBaCaL Cohort Study (ComBaCaL aHT TwiC 1 & ComBaCaL aHT TwiC 2)
Brief Title: "Community-based, eHealth Supported Management of Cardiovascular Risk Factors by Lay Village Health Workers (ComBaCaL aHT TwiC 1 & ComBaCaL aHT TwiC 2)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Agency for Development and Cooperation (SDC) (Unknown); World Diabetes Foundation (WDF) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AO_2022-00074; am22Labhardt2
Record Dates: First submitted 2023-01-02; First posted 2023-01-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Arterial Hypertension
Keywords: Community-Based Chronic Disease Care Lesotho (ComBaCaL) cohort study; low- and middle-income countries (LMICs); facility-based healthcare professionals; lay healthcare workers (LHWs); community-based aHT care models; chronic care village health workers (CC-VHWs); Lesotho Ministry of Health (MoH) Village Health Worker Program; village-based prescription; chronic care nurses (CC nurses); non-communicable diseases (NCDs); cardiovascular disease (CVD)
MeSH Terms: conditions — Hypertension; Noncommunicable Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomization for the two TwiCs will be done at cluster level, meaning that all people with aHT in one village will be offered the same care package from their local CC-VHW.
  ComBaCaL aHT TwiC 1 and aHT TwiC 2 are two cluster-randomized controlled trials that are identical in intervention, design and endpoints. They only differ in the trial population and trial hypothesis. TwiC 1 enrols individuals with uncomplicated aHT with baseline BP values above treatment targets. TwiC 2 enrols individuals with uncomplicated pharmacologically controlled aHT. In the intervention clusters community-based treatment is offered. In the control clusters participants are referred to the facility for further care after diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention villages (Active Comparator): CC-VHWs do screen, diagnosis, first-line aHT treatment for eligible participants, treatment monitoring at community-level (ComBaCaL app guides them to provide first-line antihypertensive SPCs to eligible individuals and treatment monitoring/ support to all individuals with aHT). CC- VHW offers lifestyle counselling, lipid -lowering treatment to participants with high CVD risk and antiplatelet treatment to participants with history of stroke/ myocardial infarction. Trained, supervised, mentored by chronic care nurses (CC nurses) and guided by the ComBaCaL app they follow-up persons with aHT to monitor adherence, life-style changes, treatment response, side-effects. TwiC 1: individuals with uncomplicated aHT (baseline BP above treatment targets) TwiC 2: individuals with uncomplicated pharmacologically controlled aHT. In case of complicated disease or presence of clinical alarm signs/ symptoms, participants are referred to the closest health facility for further investigation.
  Interventions: Drug: First-line antihypertensive single-pill combination (SPC)
- Control villages (Active Comparator): Control villages will follow the standard of care in the ComBaCaL cohort study. CC-VHWs will also receive tablets with the ComBaCaL app installed. They are trained, supervised and equipped to screen and diagnose aHT with subsequent referral to facility-based follow-up and care. In control villages the ComBaCaL app supports clinical decision making and documentation for screening, diagnosis and referral, but not prescription/ provision of antihypertensive or lipid-lowering medication.
  TwiC 1: enrols individuals with uncomplicated aHT with baseline BP values above treatment targets.
  TwiC 2: enrols individuals with uncomplicated pharmacologically controlled aHT.
  In case of complicated hypertension or presence of clinical alarm signs or symptoms, participants will be immediately referred to the closest health facility for further investigation.
  Interventions: Other: Standardized counselling and referral to the closest health facility

INTERVENTIONS:
Drug: First-line antihypertensive single-pill combination (SPC) — In intervention villages, participants diagnosed with aHT are offered pharmacological treatment (eHealth supported prescription of first-line antihypertensive single-pill combination (SPC)) and treatment monitoring in the villages by CC-VHWs guided by the ComBaCaL app.
  Arms: Intervention villages
Other: Standardized counselling and referral to the closest health facility — In control villages, participants diagnosed with aHT receive a standardized counselling by the CC-VHW and are referred to the closest health facility for initiation or continuation of antihypertensive treatment.
  Arms: Control villages

SUMMARY:
ComBaCaL aHT TwiC 1 and aHT TwiC 2 are two cluster-randomized controlled trials that are identical in intervention, design and endpoints. TwiC 1 enrols individuals with uncomplicated aHT with baseline BP values above treatment targets and the hypothesis is that in intervention clusters where community-based treatment is offered, a higher proportion will have controlled aHT at twelve months' follow-up as compared to control clusters where participants are referred to the facility for further care after diagnosis.

TwiC 2 enrols individuals with uncomplicated pharmacologically controlled aHT with the hypothesis that the offer of community-based antihypertensive treatment is non-inferior to facility-based care with regard to BP control rates at twelve months. The trials are nested within the ComBaCaL (Community-Based Chronic disease care Lesotho) cohort study (EKNZ ID 2022-00058, clinicaltrials.gov ID NCT05596773), a platform for the investigation of chronic diseases and their management in rural Lesotho that is maintained by local chronic care village health workers (CC-VHWs). 50% of the villages being part of the overarching ComBaCaL cohort will be randomly allocated to receive the TwiC intervention. The non-selected villages will serve as comparators and follow the regular ComBaCaL cohort activities conducted by CC-VHWs, including screening, diagnosis, standardized counselling and referral to a health facility for further therapeutic management. The TwiC intervention will be offered to all eligible people living with aHT in the sampled intervention villages. Individuals with uncomplicated uncontrolled and uncomplicated controlled aHT at baseline will be enrolled in aHT TwiC 1 and aHT 2 respectively. In case of complicated disease, unclear diagnosis, or presence of clinical alarm signs or symptoms, participants will be referred to the closest health facility for further investigation.

DETAILED DESCRIPTION:
Globally, arterial hypertension (aHT) is the single most important risk factor for early mortality. The task-shifting from facility-based healthcare professionals to lay healthcare workers (LHWs) at community-level has been identified as a promising solution to increase access to aHT treatment in low- and middle-income countries (LMICs). A cluster-randomized intervention is planned within the ComBaCaL (Community-Based Chronic disease care Lesotho) cohort study (EKNZ ID 2022-00058, clinicaltrials.gov ID NCT05596773), a platform for the investigation of chronic diseases and their management in rural Lesotho that is maintained by local chronic care village health workers (CC-VHWs). CC-VHWs are lay healthcare workers operating within the Lesotho Ministry of Health (MoH) Village Health Worker Program who receive a specific training to deliver chronic care services.

In the intervention clusters, CC-VHWs operating within the existing healthcare system will be capacitated to screen for and diagnose aHT, to prescribe first-line antihypertensive single-pill combinations (SPCs) and to monitor the treatment supported by a tailored clinical decision support application (ComBaCaL app) in their villages. The control group consists of people diagnosed with aHT living in villages that are also part of the ComBaCaL cohort but not sampled for the intervention (control villages), where CC-VHWs will only screen for and diagnose aHT with subsequent standardized counselling and referral to the closest health facility if aHT is present, but no village-based prescriptions.

The effectiveness of this intervention in two different trial populations is assessed:

* in people with uncomplicated aHT and blood pressure (BP) values above treatment target (≥ 140/90 mmHg) at baseline (aHT TwiC 1) and
* in people with uncomplicated aHT and BP values below treatment target at baseline (aHT TwiC 2).

Randomization for the two TwiCs will be done at cluster level, meaning that all people with aHT in one village will be offered the same care package from their local CC-VHW. It is planned to recruit 100 clusters (50 per study arm) for a total of 800 participants with uncontrolled aHT (TwiC 1) and 1000 participants with controlled aHT (TwiC2). 50% of the villages being part of the overarching ComBaCaL cohort will be randomly allocated to receive the TwiC intervention. The non-selected villages will serve as comparators and follow the regular ComBaCaL cohort activities conducted by CC-VHWs, including screening, diagnosis, standardized counselling and referral to a health facility for further therapeutic management. The TwiC intervention will be offered to all eligible people living with aHT in the sampled intervention villages. Individuals with uncomplicated uncontrolled and uncomplicated controlled aHT at baseline will be enrolled in aHT TwiC 1 and aHT 2 respectively. In case of complicated disease, unclear diagnosis, or presence of clinical alarm signs or symptoms, participants will be referred to the closest health facility for further investigation.

ELIGIBILITY:
Inclusion Criteria ComBaCaL-TwiC 1:

* Participant of the ComBaCaL cohort study (signed informed consent available)
* Living with aHT, defined as reporting intake of antihypertensive medication or being newly diagnosed during screening via standard diagnostic algorithm
* BP ≥140/90 mmHg at baseline

Inclusion criteria ComBaCaL-TwiC 2

* Participant of the ComBaCaL cohort study (signed informed consent available)
* Reporting intake of antihypertensive medication
* BP<140/90 mmHg at baseline

Exclusion Criteria for both ComBaCaL-TwiC 1&2:

* Reported pregnancy (at baseline or during follow-up)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1354 (Actual)
Dates: Start 2023-09-09 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure (BP) within target (<140/90 mmHg) | 12 months after enrolment
  Proportion of participants whose blood pressure (BP) is within target (<140/90 mmHg)

SECONDARY OUTCOMES:
Change in 10-year risk for a fatal or non-fatal CVD event estimated using the World Health Organization (WHO) CVD risk prediction tool | 6 and 12 months after enrolment
  The colour of the CVD risk prediction tool cell indicates the 10-year risk of a fatal or non-fatal CVD event. The value within the cell is the risk percentage. Colour coding is based on the grouping (Green<5%; Yellow5% to <10%; Red20% to <30%; Deep red≥30%)
Change in dietary habits | 6 and 12 months after enrolment
  Change in dietary habits using a shortened unquantified food frequency questionnaire adapted from an assessment tool for obesity used in South Africa
Change in International Physical Activity (PA) Questionnaire Short Form (IPAQ-SF) | 6 and 12 months after enrolment
  The IPAQ-SF addresses the number of days and time spent on PA in moderate intensity, vigorous intensity and walking of at least 10-min duration the last 7 days, and also includes time spent sitting on weekdays the last 7 days
Change in total cholesterol | 6 and 12 months after enrolment
  Change in total cholesterol
Change in abdominal circumference | 6 and 12 months after enrolment
  Change in abdominal circumference
Change in Body mass index (BMI) | 6 and 12 months after enrolment
  Change in Body mass index (BMI)
Blood pressure (BP) within target (<140/90 mmHg) | 6 months after enrolment
  Proportion of participants whose BP is within target (<140/90mmHg)
Change in mean systolic blood pressure (SBP) | 6 and 12 months after enrolment
  Mean systolic blood pressure (SBP)
Change in mean diastolic blood pressure (DBP) | 6 and 12 months after enrolment
  Mean diastolic blood pressure (DBP)
Change in occurrence of Serious Adverse Events (SAEs) | 6 and 12 months after enrolment
  Change in occurrence of Serious Adverse Events (SAEs)
Change in occurrence of Adverse Events of Special Interest (AESIs) | 6 and 12 months after enrolment
  Change in occurrence of Adverse Events of Special Interest (AESIs)
Change in proportion of participants not taking treatment at enrolment who have initiated pharmacological antihypertensive treatment | 6 and 12 months after enrolment
  Change in proportion of participants not taking treatment at enrolment who have initiated pharmacological antihypertensive treatment
Change in proportion of participants who are engaged in care | 6 and 12 months after enrolment
  Change in proportion of participants who are engaged in care (defined as reporting intake of antihypertensive medication as per prescription of a healthcare provider within the two weeks prior to assessment six and twelve months after enrolment or reaching treatment targets without intake of medication)
Change in self-reported adherence to treatment | 6 and 12 months after enrolment
  Change in self-reported adherence to treatment
Change in Quality of life (using EQ-5D-5L questionnaire) | 6 and 12 months after enrolment
  Change in Quality of life (using EQ-5D-5L questionnaire). The scale is numbered from 0 to 100. 100 means the best health you can imagine. 0 means the worst health you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Labhardt, Prof., Principal Investigator — University Hospital Basel, Division of Clinical Epidemiology; Alain Amstutz, MD, Principal Investigator — University Hospital Basel, Division of Clinical Epidemiology
Locations (2):
- SolidarMed Lesotho, Maseru, Lesotho
- University Hospital Basel, Division of Clinical Epidemiology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
* An anonymized key dataset necessary for reproducing the primary and key secondary endpoints will be made freely available in an appropriate repository, such as zenodo.org, alongside the publication of the study results. Besides removal of variables not required for key analysis, we will remove participant identifier, study site and exact date information. Requests for access to more detailed data may be made to the corresponding author by submitting a proposal, which will be reviewed by the trial consortium.
  * The statistical report for the primary and key secondary endpoints and the code to produce it will be published together with the data set.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: • Within 3 months after publication of primary results
Access Criteria: • Open access

REFERENCES:
- [Background] Gerber F, Gupta R, Lejone TI, Tahirsylaj T, Lee T, Sanchez-Samaniego G, Kohler M, Haldemann MI, Raeber F, Chitja M, Mathulise M, Kabi T, Mokaeane M, Maphenchane M, Molulela M, Khomolishoele M, Mota M, Masike S, Bane M, Sematle MP, Makabateng R, Mphunyane M, Phaaroe S, Basler DB, Kindler K, Burkard T, Briel M, Chammartin F, Labhardt ND, Amstutz A. Community-based management of arterial hypertension and cardiovascular risk factors by lay village health workers for people with controlled and uncontrolled blood pressure in rural Lesotho: joint protocol for two cluster-randomized trials within the ComBaCaL cohort study (ComBaCaL aHT Twic 1 and ComBaCaL aHT TwiC 2). Trials. 2024 Jun 6;25(1):365. doi: 10.1186/s13063-024-08226-2. PMID 38845045

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT05684055/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT05684055/SAP_001.pdf